CLINICAL TRIAL: NCT05692310
Title: Study of the Effectiveness of Central Line Placement Using an Ultraportable Ultrasound Device
Acronym: K-T-CO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-A02935-36
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Medical Imaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will have a central venous line placed using an ultraportable ultrasound device. (Experimental)
  Interventions: Other: placement of a central venous line using an ultraportable ultrasound device
- Patients will benefit from the technique of central venous line placement by conventional ultrasound (Sham Comparator)
  Interventions: Other: placing a standard central venous line

INTERVENTIONS:
Other: placing a standard central venous line — Patients will benefit from the technique of central venous line placement by conventional ultrasound.
  Arms: Patients will benefit from the technique of central venous line placement by conventional ultrasound
Other: placement of a central venous line using an ultraportable ultrasound device — Patients will have a central venous line placed using an ultraportable ultrasound device
  Arms: Patients will have a central venous line placed using an ultraportable ultrasound device.

SUMMARY:
The placement of a catheter in a large-caliber vein is sometimes necessary for the administration of treatments or the monitoring of a patient. This may be associated with complications during its realization, such as the puncture of an adjacent artery with possible formation of a hematoma or the puncture of the pleura with creation of a pneumothorax. These complications may be favored by variations in the anatomy. The use of ultrasound allows visualization of the vessels, its adjacent structures and the puncture needle along its path.

The contribution of ultrasound with the technique of venipuncture under ultrasound guidance is to date the best means of preventing complications by reducing the risk of early mechanical complications by a factor of 5 to 10 according to the studies. The retrospective, multicenter, observational study recently published by Björkander et al reported the experience of 8 Swedish hospitals with 14243 central venous catheter placements, 58% of which were in the internal jugular vein. Nearly one catheter in two was placed with the use of ultrasound (49%). One hundred and eighteen mechanical complications were recorded, of which 23 were considered serious, including 21 pneumothoraxes and 2 severe hemorrhages. Lack of ultrasound use was found to be an independent risk factor for complications in multivariate analysis by logistic regression. Despite a high level of evidence in the scientific literature on the contribution of ultrasound guidance for the placement of central venous catheters, and the recommendations of national and international learned societies published before the start of this study, almost one patient in two had not yet benefited from this technique, which could nevertheless greatly reduce the incidence of early mechanical complications.

The recent introduction of ultra-portable ultrasound scanners could encourage the generalization of the use of ultrasound, given their reduced cost. The hypothesis of the research is that the placement of a central venous catheter is similar whether the ultrasound machine is an ultra-portable ultrasound machine or a conventional ultrasound machine

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients scheduled to have a right or left jugular central venous line placed preoperatively or in the ICU .
* Patient with free, informed and express consent or emergency procedure

Exclusion Criteria:

* Absolute emergency not allowing randomization
* Pregnant woman
* Patient with suspected or proven jugular thrombosis at the insertion site
* Change of central venous line on guidewire
* Operator with no experience in central venous line placement under ultrasound
* contraindication to the placement of a jugular central venous line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
length of the procedure | 1 day
  the time in seconds between the beginning of the ultrasonographic scan after placement of the sterile protection device and the beginning of fixation of the catheter to the skin after ultrasound verification confirming its correct position.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France